CLINICAL TRIAL: NCT03026179
Title: Education of Parents About Discipline in a Way That is Culturally Sensitive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Seth Scholer, Associate Professor of Pediatrics, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PN_CultSen
Record Dates: First submitted 2015-12-09; First posted 2017-01-20 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Violence; Parenting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention parents (Other): Parents were asked to view 5-10 minutes of a program designed to educate about discipline.
  Interventions: Behavioral: Play Nicely

INTERVENTIONS:
Behavioral: Play Nicely — Play Nicely is a multimedia program that teaches parents about appropriate methods to discipline.

SUMMARY:
To determine if a brief primary care intervention can educate under-resourced and minority parents about discipline in a way that is culturally sensitive.

ELIGIBILITY:
Inclusion Criteria:

* Parents presenting with their children to a pediatric clinic.

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Cultural Sensitivity | baseline
  Parents were asked to view 5-10 minutes of an educational program. Following the clinic visit, parents were asked several questions about whether the program was culturally sensitive.

SECONDARY OUTCOMES:
Changes in discipline questionnaire | baseline
  Parents were asked if they planned to make any changes in how they discipline at home.

OTHER OUTCOMES:
Spanking questionnaire | baseline
  If parent stated that they planned to use less spanking at home, a follow up question was asked about what caused them to decide to spank less.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Scholer, MD, MPH, Principal Investigator — Vanderbilt University